CLINICAL TRIAL: NCT06218264
Title: The Role of Branched-chain Amino Acids (BCAAs) in the Stimulation of Skeletal Muscle Protein Synthesis and Glucose Uptake in Healthy Young Volunteers
Brief Title: BCAAs, Muscle Protein Synthesis and Glucose Uptake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marlou Dirks, Assistant Professor, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL82984.028.23
Record Dates: First submitted 2024-01-11; First posted 2024-01-23 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FullAA (Active Comparator): Amino acid drink containing all amino acids
  Interventions: Dietary Supplement: Ingestion of an amino acid supplement
- NoBCAA (Active Comparator): Amino acid drink containing all amino acids except for BCAAs.
  Interventions: Dietary Supplement: Ingestion of an amino acid supplement

INTERVENTIONS:
Dietary Supplement: Ingestion of an amino acid supplement — Oral intake of a supplement containing amino acids

SUMMARY:
The present study aims to quantify the insulin sensitivity and the skeletal muscle protein synthetic response to consuming a test drink containing all amino acids or all amino acids except for BCAAs.

DETAILED DESCRIPTION:
Twenty-eight healthy, young volunteers will receive a stable isotope tracer infusion (7.5h) combined with repeated blood and muscle sampling, to measure muscle protein synthesis rate in the postabsorptive state following ingestion of a drink containing all amino acids (n=14) or all amino acids except for BCAAs (n=14).

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18-35 years
* 18.5 < Body mass index < 30 kg·m2
* Recreationally active (performing non-competitive physical exercise at least one time per week for minimally 30 minutes)

Exclusion Criteria:

* Smoking
* Diabetes (Type 1, Type 2, or genetic form of diabetes)
* Any diagnosed cardiovascular (heart) disease or high blood pressure (≥140 mmHg systolic and/or ≥90 mmHg diastolic)
* Chronic use of any prescribed or over the counter pharmaceuticals (excluding oral contraceptives and contraceptive devices)
* Known allergy to lidocaine
* Regular use of dietary protein and/or amino acid supplements (>3 times per week)
* Currently involved in a structured progressive resistance training programme (>3 times per week)
* A personal or family history of thrombosis (clots), epilepsy, seizures, or schizophrenia.
* Any previous motor disorders or disorders in muscle and/or lipid metabolism
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Known severe kidney problems
* Pregnant or breastfeeding
* Unable to give consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postprandial muscle protein synthesis | 4 hours
  Muscle protein synthesis rate (FSR) prior to and following ingestion of an amino acid drink

SECONDARY OUTCOMES:
Forearm muscle glucose uptake | 7.5 hours
  Insulin sensitivity, measured as forearm glucose uptake, prior to and following ingestion of an amino acid drink
Whole-body insulin sensitivity | Four hours following ingestion of an amino acid drink
  Whole-body insulin sensitivity, calculated using a modified Matsuda index
Forearm amino acid kinetics | Prior to and for 4 hours following amino acid intake
  Plasma phenylalanine kinetics using a stable isotope tracer infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No